CLINICAL TRIAL: NCT00001566
Title: A Pilot Study of Autologous T-Cell Transplantation With Vaccine Driven Expansion of Anti-Tumor Effectors After Cytoreductive Therapy in Metastatic Pediatric Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Crystal L. Mackall, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 970052; 97-C-0052; NCT00019266 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Ewing's Sarcoma; Rhabdomyosarcoma
Keywords: Rhabdomyosarcoma; Ewing's Sarcoma; Immunotherapy; Tumor Vaccine; Interleukin-2
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma | interventions — Indinavir; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peptide vaccine/autologous T cell transplant/indinavir therapy (Experimental): Patients receive oral indinavir sulfate 350 mg/m^2 administered every 8 hours; maximum dose i.e. 800 mg every 8 hours; peptide pulsed dendritic cells 1 x 10^6 injection; harvested autologous T cells (minimum dose 1 x 10^6/kg will be thawed rapidly in 37 degree water bath and infused sequentially over 5-15 minutes.
  Interventions: Biological: therapeutic autologous dendritic cells; Drug: indinavir sulfate; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: therapeutic autologous dendritic cells — 3 syringes containing 1 x 10^6peptide pulsed dendritic cells
Drug: indinavir sulfate — Oral dose, 350 mg/m^2 administered every 8 hours. Maximum dose is 800 mg every 8 hours.
  Other Names: Crixivan
Procedure: peripheral blood stem cell transplantation — Harvested autologous T cells, minimum dose 1 x 10^6/kg will be thawed rapidly in 37 degree water bath and infused sequentially over 5-15 minutes.

SUMMARY:
This is a single arm study.

The tumor specimen is analyzed for the presence of a fusion protein which corresponds to available peptides. Patients undergo T cell harvest 10 days after an initial priming peptide-pulsed antigen presenting cell (APC) vaccine is performed.

Fresh APCs are utilized for initial priming vaccination. All subsequent vaccinations will use cryopreserved APCs. Minimum number of APCs administered per vaccination is 100,000/kg and maximum is 100,000,000/kg.

Patients undergo cytoreductive therapy for the treatment of their particular malignancy. This therapy usually consists of multiagent chemotherapy in the context of a separate protocol.

Following chemotherapy, infusion of harvested T cells followed by infusion of peptide-pulsed APC vaccinations occurs every 6 weeks for a total of 3 post-priming vaccinations. Influenza vaccine is administered by intramuscular injection concurrent to peptide-pulsed APC vaccines.

Interleukin -2 (IL-2) is administered as a continuous intravenous (IV) infusion for 4 days/week for 3 successive weeks starting on the same day as T cell /peptide-pulsed infusions.

DETAILED DESCRIPTION:
Eradication of low tumor burdens can occur in vivo when T-cell mediated responses are generated against specific tumor antigens. The Ewing's sarcoma family of tumors (ESFT) and alveolar rhabdomyosarcoma (AR) display several features which make them candidate diseases for trials of such immunotherapy. First, intensive cytotoxic chemotherapy is generally able to eradicate bulk disease in patients with metastatic disease, but tumor relapse eventually occurs in nearly all patients. Second, tumor-specific chromosomal translocations resulting in the production of novel fusion proteins have been identified in the great majority of these tumors. Peptides derived from these fusion proteins have been shown to function as tumor antigens for cytolytic T cells in animal studies. Third, studies of immune reconstitution after intensive cytotoxic therapy have provided evidence that antigen-specific T cells can be generated in vivo when the adoptive transfer of peripheral T cells and antigen are provided during the period of T cell regeneration. This process can be augmented in murine models by the use of human immunodeficiency virus (HIV) active protease inhibitor, indinavir, potentially through inhibition of programmed cell death in expanding T cells. Merging these concepts, this protocol will attempt to eradicate minimal residual disease in pediatric patients with metastatic ESFT and AR via vaccination with tumor-specific peptides undertaken concomitant with autologous T cell transplantation and indinavir.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with fusion protein bearing, metastatic malignancies of the following histologic subtypes are eligible for evaluation for treatment on this protocol: alveolar rhabdomyosarcoma (AR), and Ewing's sarcoma family of tumors (ESFT) which includes classical, atypical and extraosseous Ewing's sarcoma, peripheral primitive neuroectodermal tumors, peripheral neuroepithelioma, primitive sarcoma of bone, and ectomesenchymoma. Eligibility will not be confirmed until the presence of a tumor-specific fusion protein is documented by reverse transcription polymerase chain reaction (RT-PCR) which corresponds to one of the tumor-specific peptides available for vaccination.

Patients with Stage IV or metastatic disease are eligible to be enrolled on study at the time of initial presentation with tumor, prior to any cytoreductive therapy.

Alternatively, patients who have recurrent disease, but who have been remotely treated (completed all antineoplastic therapy greater than or equal to one year prior to enrollment for patients who are greater than 5 years of age, or completed all antineoplastic therapy greater than 6 months prior to enrollment for patients who are less than or equal to 5 years of age), are also eligible for enrollment prior to any subsequent cytoreductive therapy.

Patients who have received cytoreductive therapy for Stage IV or metastatic disease may be enrolled at the time of completion of cytoreductive therapy if an apheresis specimen is available which was collected and processed prior to cytotoxic therapy according to the guidelines described in the protocol Section 3.2.2.

Such products will have been obtained by apheresis at the Clinical Center, National Institutes of Health (NIH), with informed consent administered as per protocol 98-C-37, 97-C-0050 or as described on standard government request form 2626 for invasive procedures.

Patients must be less than or equal to 35 years at the time of initial diagnosis of alveolar rhabdomyosarcoma or ESFT, weight greater than 10 kg at the time of apheresis. Patients between 10-15 kg must be approved by the apheresis unit in the Department of Transfusion Medicine (DTM) prior to enrollment on the protocol.

All patients or their legal guardians must give written informed consent indicating their understanding of the investigational nature and risks of the study.

Patients must have adequate renal function (serum creatinine (Cr) less than 1.5 mg/dl or creatinine clearance (Cr Cl), greater than 60 ml/min./1.73 m^2 and liver function (transaminases less than 3 times normal, bilirubin less than 2.0 mg/dl). Patients will not be excluded based upon abnormal hepatic function which is related to hepatic involvement by tumor.

For remotely treated patients, a CD4 count of greater than or equal to 400 cells/mm^3 is required.

EXCLUSION CRITERIA:

Women who are pregnant or lactating.

Patients with human immunodeficiency virus infection due to confounding effects on immune function.

Patients with hepatitis B or hepatitis C infection will be excluded due to the untoward risks to personnel working with blood specimens.

Patients who require daily oral corticosteroid therapy for any underlying disease will be excluded.

Topical or inhaled corticosteroids are permitted.

Patients who are allergic to eggs, egg products, or thimerosal, or have a history of Guillain-Barre syndrome may be enrolled on study but are ineligible to receive the influenza vaccine.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 1996-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Mackall, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yanuck M, Carbone DP, Pendleton CD, Tsukui T, Winter SF, Minna JD, Berzofsky JA. A mutant p53 tumor suppressor protein is a target for peptide-induced CD8+ cytotoxic T-cells. Cancer Res. 1993 Jul 15;53(14):3257-61. PMID 7686815
- [Background] Mackall CL, Bare CV, Granger LA, Sharrow SO, Titus JA, Gress RE. Thymic-independent T cell regeneration occurs via antigen-driven expansion of peripheral T cells resulting in a repertoire that is limited in diversity and prone to skewing. J Immunol. 1996 Jun 15;156(12):4609-16. PMID 8648103
- [Background] Mackall CL, Fleisher TA, Brown MR, Andrich MP, Chen CC, Feuerstein IM, Horowitz ME, Magrath IT, Shad AT, Steinberg SM, et al. Age, thymopoiesis, and CD4+ T-lymphocyte regeneration after intensive chemotherapy. N Engl J Med. 1995 Jan 19;332(3):143-9. doi: 10.1056/NEJM199501193320303. PMID 7800006
- [Background] Zhang H, Chua KS, Guimond M, Kapoor V, Brown MV, Fleisher TA, Long LM, Bernstein D, Hill BJ, Douek DC, Berzofsky JA, Carter CS, Read EJ, Helman LJ, Mackall CL. Lymphopenia and interleukin-2 therapy alter homeostasis of CD4+CD25+ regulatory T cells. Nat Med. 2005 Nov;11(11):1238-43. doi: 10.1038/nm1312. Epub 2005 Oct 16. PMID 16227988
- [Result] Mackall CL, Rhee EH, Read EJ, Khuu HM, Leitman SF, Bernstein D, Tesso M, Long LM, Grindler D, Merino M, Kopp W, Tsokos M, Berzofsky JA, Helman LJ. A pilot study of consolidative immunotherapy in patients with high-risk pediatric sarcomas. Clin Cancer Res. 2008 Aug 1;14(15):4850-8. doi: 10.1158/1078-0432.CCR-07-4065. PMID 18676758
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-C-0052.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 patients were enrolled in this study.
Period: Overall Study
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Started | 42
Completed Immunotherapy | 23
Completed | 23
Not Completed | 19
Not completed — patients' choice to discontinue protocol | 3
Not completed — stopped after C3 due to symptomatic PD | 1
Not completed — Death | 13
Not completed — Lost to Follow-up | 1
Not completed — unable to complete initial apheresis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 18.67 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Immune Response to Tumor-specific and Non-tumor Specific Peptides During a Period of Immune Reconstitution
Description: Immune response was defined as a percent specific lysis of >10% following challenge with peptide pulsed targets, or interferon gamma production following challenge with peptide pulsed targets >2-fold that found with no-peptide controls or a proliferation index >3.0. Tumor specific peptides: Ewings sarcoma Type 1: EF-1 (EWS/FLI-1)*SSSYGQQN/PSYDSVRRGA,Ewing's Sarcoma Type 2: EF-2 (EWS/FLI-2)* SSSYGQ/QSSLLAYNT, Alveolar rhabdomyosarcoma: PXFK (PAX3/FKHR)† TIGNGLSPQ/NSIRHNLSL. Non-tumor specific peptide:HPV16E7 MLDLQPETT-MET-9-THR. See protocol link module for additional information re: peptides.
Time Frame: 20 weeks post vaccination
Measure: Number; unit: Participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 23
Participants
  Immune response to tumor specific peptides | 9
  Immune response to non-tumor specific peptides | 23

2. Primary Outcome: The Percent of Patients Who Recover CD4 Counts Within 6 Months of Completion of Chemotherapy
Description: CD4 counts were measured from peripheral blood using standard flow cytometric techniques at the following timepoints: 2 months post-chemotherapy, 4 months post-chemotherapy and 6 months post-chemotherapy. To be eligible for evaluation for this endpoint, patient much have been <10 years of age and sustained a CD4 count of <300 cells/mcl upon completion of standard therapy. Recovery was defined as a CD4 count > 500 cells/mcl at any timepoint within 6 months of completing chemotherapy.
Time Frame: 2 to 6 months
Measure: Number; unit: Percentage of participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 16
Percentage of participants | 12.5

3. Primary Outcome: Number of Participants With an Immune Response to the Translocation Breakpoint Peptide
Description: Immune responses were measured following 3 sequential influenza vaccines during the same period as the peptide-pulsed dendritic cell vaccines.
Time Frame: 5 years
Measure: Number; unit: Participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 23
Participants | 9

4. Secondary Outcome: Percentage of Participants Overall Survival
Description: Overall survival is defined as the time between the first day of treatment to the day of death.
Time Frame: 5 years
Measure: Number; unit: Percentage of participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 42
Percentage of participants | 43

5. Secondary Outcome: Percent of Participants: Event Free Survival
Description: Event free survival is calculated from the date of diagnosis for patients enrolled with newly diagnosed metastatic disease and from the date of the last recurrence detection before enrollment on this study for patients with recurrent disease.
Time Frame: 5 years
Measure: Number; unit: Percentage of participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 42
Percentage of participants | 31

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 5 years
Measure: Number; unit: Participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 42
Participants | 27

7. Primary Outcome: Number of Participants With an Immune Response to Non-Tumor-specific Peptide E7
Description: Immune response was defined as a percent specific lysis of >10% following challenge with peptide pulsed targets, or interferon gamma production following challenge with peptide pulsed targets >2-fold that found with no-peptide controls or a proliferation index >3.0.
Time Frame: 5 years
Population: 12 patients were human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2+) and therefore evaluable for response to E7 peptides.
Measure: Number; unit: Participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 12
Participants | 3

8. Primary Outcome: Number of Participants With an Immune Response to Tumor-Specific Peptides at the Time of Presentation
Description: Immune response was defined as a percent specific lysis of >10% following challenge with tumor peptide pulsed targets, or interferon gamma production following challenge with tumor peptide pulsed targets >2-fold that found with no-peptide controls or a proliferation index >3.0 to tumor peptide targets.Tumor specific peptides: Ewings sarcoma Type 1: EF-1 (EWS/FLI-1)*SSSYGQQN/PSYDSVRRGA,Ewing's Sarcoma Type 2: EF-2 (EWS/FLI-2)* SSSYGQ/QSSLLAYNT, Alveolar rhabdomyosarcoma: PXFK (PAX3/FKHR)† TIGNGLSPQ/NSIRHNLSL. See protocol link module for additional information re: peptides.
Time Frame: Once per enrollment
Measure: Number; unit: Participants
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 23
Participants | 5

9. Secondary Outcome: Median Overall Survival
Description: Overall survival is defined as the time between the first day of treatment to the day of death.
Time Frame: 5.4 years
Measure: Median (Full Range); unit: Years
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Number analyzed (Participants) | 42
Years | 4.1 [3.4 to 5.4]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy
Serious Adverse Events (participants affected / at risk) | 15/42
Other Adverse Events (participants affected / at risk) | 27/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy (N=42)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
CPK (Creatine phosphokinase) (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
DVT (deep vein thrombosis) (Vascular disorders) | 1 (1)
Elevated total bilirubin (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (Investigations) | 1 (2)
Neutropenia (Investigations) | 3 (4)
Neutrophils (Investigations) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Rash with macules/papules (Skin and subcutaneous tissue disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peptide Vaccine/Autologous T Cell Transplant/Indinavir Therapy (N=42)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (5)
Achiness (Musculoskeletal and connective tissue disorders) | 1 (1)
Achy (General disorders) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 1 (6)
Acne (rash) on chest (Skin and subcutaneous tissue disorders) | 1 (4)
Alkaline phosphate elevated (Metabolism and nutrition disorders) | 7 (10)
ALT (SGPT) (Metabolism and nutrition disorders) | 1 (5)
Anemia (Blood and lymphatic system disorders) | 6 (9)
Anxiety (Psychiatric disorders) | 2 (2)
Anxiety symptoms (Psychiatric disorders) | 1 (1)
AST (SGOT) (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Bad taste in mouth (Gastrointestinal disorders) | 1 (1)
Bilateral flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bitter taste in mouth (Gastrointestinal disorders) | 1 (4)
Bruise (Injury, poisoning and procedural complications) | 1 (1)
Chelitis (Gastrointestinal disorders) | 1 (1)
Chest tightness (General disorders) | 1 (1)
Chills (General disorders) | 7 (14)
Cold (General disorders) | 2 (2)
Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Cough (dry) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (mild, intermittent) (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Cough nonproductive (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cranky (General disorders) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 3 (4)
Decreased flexibility swelling left leg (General disorders) | 1 (1)
Decreased uric acid (Metabolism and nutrition disorders) | 1 (1)
Decreased urine output (o/p) (Renal and urinary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Discoloration skin (L) hand (Skin and subcutaneous tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dizzy (Nervous system disorders) | 1 (1)
Double vision (Eye disorders) | 1 (1)
Drainage on foot (Musculoskeletal and connective tissue disorders) | 1 (2)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry heaves (Gastrointestinal disorders) | 1 (1)
Dry lips (Gastrointestinal disorders) | 2 (2)
Dry scaly peeling skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dry scaly skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5)
Ear pain/infection (Ear and labyrinth disorders) | 1 (1)
Ears ringing (Ear and labyrinth disorders) | 1 (4)
Ears ringing and clogged (Ear and labyrinth disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Edema media R mid-thigh (General disorders) | 1 (1)
Edema on foot (General disorders) | 1 (2)
Edema, facial (General disorders) | 2 (2)
Elevated creat (Investigations) | 1 (1)
Elevated creatin (Investigations) | 1 (1)
Elevated D bili (Hepatobiliary disorders) | 4 (4)
Elevated glucose (Metabolism and nutrition disorders) | 2 (2)
Elevated LFT's (liver function tests) (Hepatobiliary disorders) | 1 (1)
Elevated magnesium (Metabolism and nutrition disorders) | 2 (3)
Elevated SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 8 (8)
Elevated SGPT (serum glutamic pyruvic transaminase) (Investigations) | 10 (14)
Elevated BUN (Investigations) | 1 (1)
Elevated creatinine (Investigations) | 1 (1)
Emesis (Gastrointestinal disorders) | 2 (7)
Eosinophilia (Investigations) | 13 (33)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Eye pain (Eye disorders) | 1 (1)
Eye swollen (Eye disorders) | 1 (1)
Eyes watery (Eye disorders) | 1 (1)
Fatigue (General disorders) | 16 (24)
Fever (General disorders) | 12 (25)
Fever (by touch) (General disorders) | 1 (1)
Fever (by touch-low grade) (General disorders) | 1 (1)
Fever blister (General disorders) | 1 (3)
Fever-low grade (by touch) (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
flu symptoms (General disorders) | 3 (8)
Flu-like symptoms (General disorders) | 4 (4)
Flush cheeks (General disorders) | 1 (1)
Flush, facial (General disorders) | 2 (2)
Flushed (General disorders) | 1 (1)
Flushed skin (General disorders) | 1 (1)
Flushing (General disorders) | 2 (3)
Foot drop (General disorders) | 1 (1)
Gas build-up (Gastrointestinal disorders) | 1 (1)
Gas pains (Gastrointestinal disorders) | 1 (1)
Generalized pain (General disorders) | 1 (1)
Glands swoll (General disorders) | 1 (1)
Glucosuria (Metabolism and nutrition disorders) | 1 (1)
Gum line bump (L. upper) (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 11 (14)
Heartburn (Gastrointestinal disorders) | 2 (7)
Hematuria (Renal and urinary disorders) | 7 (10)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage sclera (Eye disorders) | 1 (1)
Hives (Skin and subcutaneous tissue disorders) | 1 (1)
Hot feeling (Vascular disorders) | 1 (1)
Hyperbilirubin (Hepatobiliary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (2)
Hyperthyroid (Endocrine disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 4 (4)
Hypothyroid (Endocrine disorders) | 2 (2)
Impetigo (Skin and subcutaneous tissue disorders) | 1 (1)
INC SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 1 (2)
INC SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (5)
Increase fatigue (General disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Induration (Skin and subcutaneous tissue disorders) | 1 (2)
Induration injection site (Skin and subcutaneous tissue disorders) | 1 (5)
Inf IV site (Infections and infestations) | 1 (1)
Injection sclera (Eye disorders) | 1 (1)
Injection reaction (General disorders) | 7 (38)
Insomnia (Psychiatric disorders) | 3 (4)
Intermittent pain in shaft of R tibia (Musculoskeletal and connective tissue disorders) | 3 (3)
Intermittent H/A (headache) (Nervous system disorders) | 3 (6)
Intermittent cramping legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Intermittent fatigue (General disorders) | 1 (4)
Intermittent insomnia (Psychiatric disorders) | 1 (3)
Irritable (General disorders) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 1 (1)
Itching (chest) (Skin and subcutaneous tissue disorders) | 1 (1)
Itching/injection site (Skin and subcutaneous tissue disorders) | 1 (3)
Itchy L. leg (Skin and subcutaneous tissue disorders) | 1 (1)
Itchy scratch under left eye (Skin and subcutaneous tissue disorders) | 1 (1)
Jaw pain (General disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Kidney stone (Renal and urinary disorders) | 1 (1)
L anterior chest pain (General disorders) | 1 (1)
Left chest pressure (General disorders) | 1 (1)
Left ear ringing (Ear and labyrinth disorders) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Lethargic (Nervous system disorders) | 1 (1)
Leukocytes (Investigations) | 1 (7)
Lips numb (Nervous system disorders) | 2 (2)
Loose stool (Gastrointestinal disorders) | 2 (8)
Loose stools (Gastrointestinal disorders) | 1 (1)
Loss of balance (Ear and labyrinth disorders) | 1 (1)
Low albumin (Metabolism and nutrition disorders) | 3 (3)
Low CO2 (Investigations) | 1 (1)
Low potassium (Metabolism and nutrition disorders) | 1 (1)
Lower back soreness (Musculoskeletal and connective tissue disorders) | 2 (3)
Malaise (General disorders) | 5 (6)
Malleolus (pain) (General disorders) | 1 (1)
Minor sore throat (Gastrointestinal disorders) | 1 (1)
Muscle aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia-bilateral thighs (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 (18)
Nasal drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (24)
Nausea/vomiting (Gastrointestinal disorders) | 2 (2)
Neutropenia (Investigations) | 5 (6)
Neutrophils (Investigations) | 1 (5)
Night sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nose congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Numbness in feet and hands (Nervous system disorders) | 2 (3)
Occipital (mild pain) (Nervous system disorders) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain injection site (General disorders) | 1 (1)
Pain R foot (General disorders) | 1 (1)
Pain R hip (General disorders) | 1 (1)
Pain tailbone (General disorders) | 1 (2)
Patchy dry skin/itch trunk (Skin and subcutaneous tissue disorders) | 1 (2)
Perior edema (General disorders) | 1 (2)
Petechiae (Blood and lymphatic system disorders) | 1 (1)
Platelets (Investigations) | 1 (2)
Pressure in chest with inhalation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pretib edema (General disorders) | 1 (1)
Prickling sensation (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 8 (17)
Pruritis (Skin and subcutaneous tissue disorders) | 3 (3)
Ptosis (Eye disorders) | 1 (1)
Puffy face (General disorders) | 1 (1)
Quad muscle soreness (Musculoskeletal and connective tissue disorders) | 1 (4)
Quad/muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Rash, chest (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, arm/chs (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/redness (top of arm) (Skin and subcutaneous tissue disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scrape on face (Injury, poisoning and procedural complications) | 1 (1)
Scratch under left eye (Injury, poisoning and procedural complications) | 1 (1)
Shoulder pain (General disorders) | 1 (2)
Skin peeling (Skin and subcutaneous tissue disorders) | 1 (1)
Skin sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Sore mouth (Gastrointestinal disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Soreness under ribs (Musculoskeletal and connective tissue disorders) | 1 (1)
Soreness/achiness (Musculoskeletal and connective tissue disorders) | 1 (1)
Stiff neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomach ache (Gastrointestinal disorders) | 3 (4)
Stomach burning (Gastrointestinal disorders) | 1 (3)
Stomach pain (Gastrointestinal disorders) | 3 (3)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stye (L) lower corner eye (Eye disorders) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Swell ankle (General disorders) | 1 (1)
Swell tongue (General disorders) | 1 (1)
Swelling lip (General disorders) | 1 (1)
Swelling-lower extremity (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (9)
Tiredness (General disorders) | 1 (1)
Ulceration (R) heel (Skin and subcutaneous tissue disorders) | 1 (4)
Ulceration L heel (Skin and subcutaneous tissue disorders) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 3 (3)
URI (upper respiratory infection) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Vascular (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (15)
Weakness (General disorders) | 1 (1)
Weakness (L. leg) (Musculoskeletal and connective tissue disorders) | 1 (2)
Weight gain (Investigations) | 6 (6)
Weight loss (Investigations) | 3 (3)
Decreased L leg flexibility (General disorders) | 2 (2)
Elevated uric acid (Metabolism and nutrition disorders) | 1 (1)
Elev phos (Metabolism and nutrition disorders) | 1 (1)
Itchy legs (Skin and subcutaneous tissue disorders) | 1 (4)
Pain, legs (General disorders) | 1 (1)
Elevated total bilirubin (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No